CLINICAL TRIAL: NCT07284836
Title: Phase II Trial of Albumin-Bound Paclitaxel Combined With Nedaplatin (TP) Via Hepatic Arterial Infusion for Advanced Breast Cancer Patients With Liver Metastases After Failure of Standard Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Hu Hai, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2024-467
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Hepatic Artery Infusion; Liver Metastasis of Breast Cancer
MeSH Terms: interventions — Albumin-Bound Paclitaxel; nedaplatin

STUDY DESIGN:
Intervention Model Description: Intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abraxane+Nedaplatin (Experimental): 1. Abraxane：Dosage: 200 mg，Route of Administration: Via hepatic arterial catheter infusion，Frequency: Every three weeks，Infusion Duration: Approximately 30 minutes
  2. Nedaplatin：Dosage: 100 mg，Route of Administration: Via hepatic arterial catheter infusion，Frequency: Every three weeks，Infusion Duration: Approximately 30 minutes，Treatment Cycle: Each cycle spans 3 weeks, for a total of 6-8 cycles. The exact number of cycles may be adjusted based on the patient's tolerance and disease response.
  Interventions: Drug: Abraxane; Drug: Nedaplatin

INTERVENTIONS:
Drug: Abraxane — Abraxane，200 mg，Via hepatic arterial catheter infusion，Every three weeks
Drug: Nedaplatin — Nedaplatin，100 mg，Via hepatic arterial catheter infusion，Every three weeks

SUMMARY:
Study Objective: To Evaluate the Efficacy of Albumin-Bound Paclitaxel Combined with Nedaplatin via Hepatic Arterial Infusion as Later-Line Therapy for Breast Cancer Patients with Liver Metastases After Failure of Standard Treatment.

Outcome Measures：Primary Outcome: Liver Progression-Free Survival (LPFS) Secondary Outcomes:Liver Objective Response Rate (LORR)、Progression-Free Survival (PFS) and Overall Survival (OS)

Participants will:

* Albumin-bound paclitaxel + nedaplatin (TP) regimen is administered via hepatic arterial infusion chemotherapy on Day 1 of each cycle.
* Tumor response will be assessed every 6 weeks (±7 days) according to RECIST 1.1 criteria until disease progression is determined by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver metastases from breast cancer pathologically confirmed via surgery or biopsy.

  * Advanced breast cancer patients with imaging-confirmed visceral tumor burden solely confined to liver metastases.

    * Patients who have previously failed at least two lines of standard therapy (including endocrine therapy, chemotherapy, or targeted therapy), or those for whom researchers determine that local therapy would yield greater benefit.

      * Age 18-70 years.

        * ECOG (Eastern Cooperative Oncology Group) performance status score of 0-2. • 0: Fully active, without any restrictions; • 1: Restricted in physically strenuous activity but ambulatory and able to carry out light work; • 2: Ambulatory and capable of all self-care but unable to carry out any work activities.

          * Liver function score (e.g., Child-Pugh) Class A-B.

            • Class A (5-6 points): Good hepatic reserve, well tolerated to surgery, low incidence of postoperative complications and mortality;

            • Class B (7-9 points): Moderately impaired hepatic reserve, poorly tolerated to surgery, increased postoperative complications and mortality;

            • Class C (≥10 points): Severely impaired hepatic reserve, very poorly tolerated to surgery, high risk of postoperative complications and mortality; surgery is generally not recommended.

            ⑦ Adequate organ function.

            • Hemoglobin ≥90 g/L, white blood cells ≥3.5×10⁹/L, neutrophils ≥1.5×10⁹/L, platelets ≥100×10⁹/L;

            • Serum creatinine ≤1.0×upper normal limit (UNL), and creatinine clearance >60 mL/min;

            • Alanine aminotransferase (ALT) ≤1.5×UNL, aspartate aminotransferase (AST) ≤1.5×UNL, alkaline phosphatase (ALP) ≤1.5×UNL;

            • Total bilirubin (TBIL) ≤1.5×UNL;

            • No severe abnormalities on electrocardiogram, left ventricular ejection fraction (LVEF) ≥50%;

            • Absence of other severe medical conditions or comorbidities that would preclude tolerance to the clinical trial intervention.
            * Signed informed consent, indicating understanding of the trial's purpose, risks, and potential benefits.

Exclusion Criteria:

1. History of other malignancies.
2. Breast and chest wall recurrence, brain metastases, multiple bone metastases with fracture risk, or visceral metastases outside the liver.
3. Tumor volume ≥70% of liver volume.
4. History of heart failure (NYHA class >I), myocardial infarction, unstable angina, stroke, or poorly controlled arrhythmia.
5. Active infection, severe allergic reactions, or autoimmune diseases, including but not limited to:

   * Active tuberculosis (TB), currently receiving or having received anti-TB treatment within the past year;
   * HIV infection (HIV1/2 antibody positive);
   * Active hepatitis B or hepatitis C virus infection;
   * History of systemic lupus erythematosus, rheumatoid arthritis, chronic lymphocytic thyroiditis, hyperthyroidism, polyarteritis nodosa, autoimmune hemolytic anemia, etc.
6. Administration of live attenuated vaccines within 4 weeks prior to enrollment or planned during the study period.
7. Uncontrolled hypertension, diabetes, or other serious diseases.
8. Severe uncontrolled dysfunction of the liver, kidneys, lungs, or other vital organs.
9. Pregnant or lactating patients.
10. History of mental illness.
11. Known allergy to albumin-bound paclitaxel, nedaplatin, or related drugs.
12. Current participation in another clinical trial.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Liver progression-free survival, L-PFS | Up to approximately 33 months
  The period from the first liver artery chemotherapy infusion to the time of the first recorded liver tumor progression or the patient's death

SECONDARY OUTCOMES:
Liver objective response rate, L-ORR | Up to approximately 33 months
  The proportion of patients in the treatment group who achieved complete response (CR) or partial response (PR) for liver masses.
progression-free survival, PFS | Up to approximately 33 months
  From the time of the first hepatic artery chemotherapy infusion to the time of the first recorded local tumor progression or the patient's death
overall survival, OS | The time from date of enrollment to the date of death due to any cause up to approximately 33 months
  overall survival, OS

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided